CLINICAL TRIAL: NCT02107118
Title: H-34570: PHASE I Study: The Use of Autologous Adipose Tissue-Derived Mesenchymal Stem Cell (AdMSC) for the Improvement of Erectile and Cardiac Function in Aging Men
Brief Title: Stem Cells for the Improvement of Erectile and Cardiac Function in Aging Men
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Contract issues
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohit Khera, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-34570 No.11-13-40-07
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Erectile Dysfunction; Cardiac Disease
Keywords: Stem cells; cardiovascular disease; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM 1: AdMSC: adipose stem cells (Active Comparator): AdMSC: Autologous adipose tissue-derived mesenchymal stem cell. Adipose tissue will be harvested from all patients as previously described and stem cells will be cultured.
  Interventions: Biological: ARM 1: AdMSC: adipose stem cells
- ARM 2 Placebo (Placebo Comparator): Adipose tissue will be harvested from all patients as previously described and stem cells will be cultured. For those subjects in the placebo arm, the stem cells will be frozen for later use after one year when the patients cross over into the treatment arm.
  Interventions: Other: ARM 2: Placebo

INTERVENTIONS:
Biological: ARM 1: AdMSC: adipose stem cells — Adipose tissue will be harvested from all patients as previously described and stem cells will be cultured. Cells are returned to the study doctor for installation into the subject every 2 weeks for 3 months.
  Other Names: ARM 1: AdMSC: Adipose derived mesenchymal stem cells
  Arms: ARM 1: AdMSC: adipose stem cells
Other: ARM 2: Placebo — Adipose tissue will be harvested from all patients as previously described and stem cells will be cultured. For those subjects in the placebo arm, the stem cells will be frozen for later use after one year when the patients cross over into the treatment arm.
  Other Names: ARM 2 Placebo
  Arms: ARM 2 Placebo

SUMMARY:
Men who present with erectile dysfunction as defined as an IIEF (International Index of Erectile Function) score less than 21 will be evaluated for risk factors for cardiovascular disease (CVD). This is a single-blind study. Subjects will be randomized in a 2:1 fashion for treatment (ARM 1) versus placebo (ARM 2). Adipose tissue (fat) will be harvested from all patients and stem cells will be cultured. For those patients in the placebo arm the stem cells will be frozen for later use after one year when the patients cross over into the treatment arm.

DETAILED DESCRIPTION:
Baseline assessment of patients will include completion of 6 questionnaires, EKG (electrocardiogram), vision testing using a standard eye chart, markers of endothelial dysfunction hormone evaluation, laboratory blood tests, vital signs, penile ultrasound (optional), echocardiogram, chest x-ray, and endothelial function assessment (Endopat).

The adipose tissue sample is sent to Celltex's state-of-the-art laboratory in Houston, Texas. For those subjects in the placebo arm, the stem cells will be frozen for later use after one year when the patients cross over into the treatment arm. The subject (patient) will receive an infusion of either autologous stem cells (cells made from his own fat tissue) or placebo every 2 weeks for 3 months. Placebo will be in the form of normal saline. Subjects will be closely monitored every two weeks for first 3 months and once the treatment is complete, subjects will be monitored every 3 months for the first year. Each of the previously mentioned tests will be performed at the 3, 6, 9, and 12 month mark. However, the penile ultrasound (optional) and the echocardiogram will be performed only at the 3 and 12 month mark.

ELIGIBILITY:
Inclusion Criteria:

* Men 40 years of age or older
* Men with erectile dysfunction as defined by IIEF score less than 21
* Men with endothelial dysfunction as defined as an RHI score less than 2
* Men with normal testosterone levels (300 ng/dl)

Exclusion Criteria:

* Men under the age of 40
* Men with normal erectile function
* Men with normal endothelial function
* Men with low testosterone levels (less than 300ng/dl)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2020-03 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Improvements in IIEF scores of greater than 2 | 12 months
  The analysis will allow us to assess if stem cells can improve IIEF scores. The IIEF will be given at the 3, 6, 9, and 12 month visits.

SECONDARY OUTCOMES:
Improvements in RHI (reactive hyperemic index) scores of greater than 0.3 | 12 months
  The analysis will allow us to assess if stem cells can improve endothelial function. The RHI scores will be reviewed at the 3, 6, 9, and 12 month visits.

OTHER OUTCOMES:
Improvements in penile duplex | 12 months
  The analysis will allow us to assess if stem cells can improve penile duplex. The penile duplex will be given at the 3 and 12 month visits.
Improvements in echocardiogram | 12 months
  The analysis will allow us to assess if stem cells can improvement results of the echocardiogram. The echocardiogram will be done at the 3 and 12 month visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Khera, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Khera M, Albersen M, Mulhall JP. Mesenchymal stem cell therapy for the treatment of erectile dysfunction. J Sex Med. 2015 May;12(5):1105-6. doi: 10.1111/jsm.12871. No abstract available. PMID 25974235